CLINICAL TRIAL: NCT02891239
Title: Clinical Study to Evaluate the Performance of the PicoWay 1064 nm/ 785 nm/ 532nm Picosecond Laser for Treatment of Benign Pigmented Lesions
Brief Title: 785nm Picosecond Laser for Treatment of Benign Pigmented Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Syneron Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DHF21261
Record Dates: First submitted 2016-09-01; First posted 2016-09-07 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Benign Pigmented Lesions
Keywords: laser treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PicoWay laser treatment (Experimental): 3 wavelength tattoo treatment with picosecond laser (PicoWay)
  Interventions: Device: PicoWay

INTERVENTIONS:
Device: PicoWay — solid state laser capable of delivering energy at wavelengths of 1064 nm or 532 nm or wavelength of 785 nm that was added to the system
  Other Names: PicoWay device

SUMMARY:
This is an open-label, multi-center study. Subjects in this study will receive up to eight (8) treatments in 11±5 weeks (6-16 weeks) interval, with the PicoWay device using the 785 nm wavelength alone or combined with 1064 nm or 532 nm wavelengths. Subjects will return for one follow-up (FU) visit at the clinic at 8 weeks following the last treatment.

DETAILED DESCRIPTION:
This study is a prospective clinical study to demonstrate the safety and efficacy of the PicoWay device for benign pigmented lesion treatment.

Up to a total of 60 healthy candidates, who are seeking treatment/clearance of benign pigmented lesions, will be enrolled at up to 3 participating study sites. Subjects will receive up to eight (8) PicoWay treatments at 11±5 (6-16) week's intervals. Prior to each consecutive treatment, the investigator will decide, based on degree of clearance assessment, should the subject undergo additional treatment or proceed to the 8-weeks follow-up (FU) visit with no more treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy female and male subjects between 18 to 70 years of age
2. Fitzpatrick skin type I-VI
3. Presence of unwanted benign pigmented lesions including but not limited to solar lentigines, freckles, café au lait, melasma, Nevis of Ota, Nevus of Ito and hyperpigmentation. Multiple lesions can be treated.
4. Willing to receive the proposed PicoWay treatments and comply with all study (protocol) requirements to remove unwanted benign pigmented lesions.
5. Willing to have photographs and images taken of the treated areas to be used in evaluations, publications and presentations (subject identity will be masked).
6. For female subjects: not pregnant or lactating and is either post-menopausal, surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment (i.e., oral contraceptives, contraceptive implant, barrier methods with spermicide or abstinence)
7. Informed consent process is completed and subject consent is signed.

Exclusion Criteria:

1. Pregnant or planning to become pregnant, having given birth less than 3 months ago, and/or breast feeding
2. Hypersensitivity to light exposure
3. Taking medication(s) for which sunlight is a contraindication
4. Active sun tan
5. Suffering from significant skin conditions in the treated areas or inflammatory skin conditions, including, but not limited to, open lacerations or abrasions, hidradenitis, or dermatitis of the treatment area prior to treatment (duration of resolution as per the Investigator's discretion) or during the treatment course
6. History of squamous cell carcinoma or melanoma
7. History of keloid scarring, abnormal wound healing and / or prone to bruising
8. Use of oral isotretinoin (Accutane®) within 12 months of initial treatment or plans on using during the course of the study. Note: Skin must regain its normal degree of moisture prior to treatment, e.g., lack of noticeable skin flaking, skin peeling and skin surface roughness
9. History of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or currently using immunosuppressive medications
10. Known allergy to lidocaine, tetracaine, Xylocaine or epinephrine
11. Has had a laser procedure, a peel or has used lightening creams in the area to be treated with in the past six months
12. Subjects with pigmented lesions that are considered not acceptable by the study doctor or any condition that, in the study doctor's opinion, would make it unsafe to treat
13. As per the investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Blinded evaluation of pigmentation clearance | 8 weeks post final treatment
  Global percentage of pigmentation clearance, as assessed by blinded evaluators based on comparing pre and post treatment photos.

SECONDARY OUTCOMES:
Global percentage of pigmentation clearance | 8 weeks post final treatment
  Global percentage of pigmentation clearance, as assessed by study investigators based on comparing pre and post treatment photos.
Number of patients with adverse events | Through study completion, average of 1 year
  Based on rate and severity of treatments with the PicoWay laser treatment
Investigator satisfaction with treatment | 8 weeks post final treatment
  A 5-point satisfaction scale will be used by study investigators to assess satisfaction with treatment outcome
Subject satisfaction with treatment | 8 weeks post final treatment
  A 5-point satisfaction scale will be used by subjects to assess satisfaction with treatment outcome

CONTACTS AND LOCATIONS:
Overall Officials: Konika Schallen, MD, Principal Investigator — Syneron Candela Institute for Education Clinic
Locations (1):
- Syneron Candela Institute for Education Clinic, Wayland, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bernstein EF, Schomacker KT, Basilavecchio LD, Plugis JM, Bhawalkar JD. A novel dual-wavelength, Nd:YAG, picosecond-domain laser safely and effectively removes multicolor tattoos. Lasers Surg Med. 2015 Sep;47(7):542-548. doi: 10.1002/lsm.22391. Epub 2015 Jul 14. PMID 26175187
- [Background] Levin MK, Ng E, Bae YS, Brauer JA, Geronemus RG. Treatment of pigmentary disorders in patients with skin of color with a novel 755 nm picosecond, Q-switched ruby, and Q-switched Nd:YAG nanosecond lasers: A retrospective photographic review. Lasers Surg Med. 2016 Feb;48(2):181-7. doi: 10.1002/lsm.22454. PMID 26922302